CLINICAL TRIAL: NCT01068132
Title: Prognostic Factors for Patients With Advanced Colorectal Cancer Treated With Cetuximab. An Italian Trial
Brief Title: Prognostic Factors for Patients With Advanced Colorectal Cancer Treated With Cetuximab.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regione Lombardia (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Istituto Clinico Humanitas (Other); A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-007524-25
Record Dates: First submitted 2009-05-04; First posted 2010-02-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; KRAS; PTEN
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cetuximab+FOLFIRI: cetuximab 500 mg/ m² starting dose, following everytwo- week doses of 500 mg/ m², given d1, followed after 1 hour by FOLFIRI: irinotecan 180 mg/m2 on day 1 with LV 100 mg/m2 administered as a 2-hour infusion before FU 400 mg/m2 administered as an intravenous bolus injection, and FU 600 mg/m2 as a 22-hour infusion immediately after FU bolus injection on days 1 and 2
  Interventions: Drug: Cetuximab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab — cetuximab 500 mg/ m² starting dose, following everytwo- week doses of 500 mg/ m², given d1,
Drug: FOLFIRI — irinotecan 180 mg/m2 on day 1 with LV 100 mg/m2 administered as a 2-hour infusion before FU 400 mg/m2 administered as an intravenous bolus injection, and FU 600 mg/m2 as a 22-hour infusion immediately after FU bolus injection on days 1 and 2

SUMMARY:
Italian, multicentre, non comparative trial in patients with advanced Colorectal Cancer(CRC)and KRAS wild-type, defined by molecular evaluation.

Patients will receive Cetuximab + FOLFIRI until disease progression, unacceptable toxicity developed or patient refusal.

The aim of this study is to assess the prognostic role of PTEN in terms of Progression free survival.

Although the role of Cetuximab as first line treatment in metastatic CRC will be soon established, it is still unclear which is the best schedule for Cetuximab and the role of biological factors in order to select the most appropriate subset of pts for recommending Cetuximab. The data supporting a benefit of Cetuximab in KRAS wild-type pts open the perspective to study the role of other molecular markers in this subset of pts.

On the basis of these considerations this study is aimed at testing a different schedule of Cetuximab and better characterize the prognosis of pts for which Cetuximab is appropriate.

DETAILED DESCRIPTION:
Pts meeting eligibility criteria will be registered, providing the availability of material for molecular analysis. Tumour specimens and blood sample will be collected to perform genomic, ICH and proteomic analyses in order to identify the molecular characteristics of tumour.

After the availability of KRAS evaluation, only the data of KRAS wild-type pts will be collected.

Access to registration system will be allowed via web.

Patients,KRAS wild-type receive:

- Cetuximab+FOLFIRI: cetuximab 500 mg/ m² starting dose, following everytwo- week doses of 500 mg/ m², given d1, followed after 1 hour by FOLFIRI: irinotecan 180 mg/m2 on day 1 with LV 100 mg/m2 administered as a 2-hour infusion before FU 400 mg/m2 administered as an intravenous bolus injection, and FU 600 mg/m2 as a 22-hour infusion immediately after FU bolus injection on days 1 and 2

ELIGIBILITY:
Inclusion criteria

* Signed written informed consent for biological analysis (all pts)
* Signed written informed consent for enrolment (pts with KRAS wild type)
* Male or female aged > or = 18 years
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* KRAS evaluation availability with wild-type result
* Metastatic CRC not suitable for curative-intent resection
* Availability of tumour samples (or able and willing to provide tumour sample) and blood for biological analysis
* Presence of at least one lesion measurable unidimensionally by computed tomography (CT) scan or magnetic resonance imaging (MRI). (index lesion(s) must not lie within an irradiated area)
* Eastern cooperative oncology group-performance status (ECOG-PS) <2

Exclusion criteria

* Brain metastasis (known or suspected)
* Previous chemotherapy for metastatic CRC (any). Adjuvant therapy is allowed if the chemotherapy treatment free interval is > 6 months
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to study entry
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to entry
* Previous exposure to HER-axis -pathway targeting therapy
* Leucocytes <3.0 x 109/L and neutrophils <1.5 x 109/L, platelets <100 x 109/L, and hemoglobin <9 g/dL
* Bilirubin level either normal or >1.5 x ULN
* ASAT and ALAT >2.5 x ULN (>5 x ULN if liver metastasis are present)
* Serum creatinine >1.5 x ULN
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Pre-existing neuropathy > grade 1
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Pts with a previous malignancy but without evidence of disease for > or equal 5 years will be allowed to enter the trial)
* Pregnancy or lactation
* Inadequate contraception (male or female pts) if of childbearing or procreational potential
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | untill 48 months

SECONDARY OUTCOMES:
Overall survival | untill 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Labianca, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (7):
- Italy (7):
  - Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - Ospedale di Treviglio e Caravaggio, Treviglio, Bergamo
  - IRCCS San Raffaele, Milan, Milano
  - Istututo Clinico Humanitas, Rozzano, Milano
  - Ospedale Morelli Sondalo, Sondalo, Sondrio
  - Ospedale di Sondrio, Sondrio, Sondrio
  - Ospedale di Saronno, Saronno, Varese